CLINICAL TRIAL: NCT04798339
Title: A Phase 1b/2 Study Evaluating the Safety and Efficacy of Canakinumab With Darbepoetin Alfa in Patients With Lower-Risk Myelodysplastic Syndromes (MDS) Who Have Failed Erythropoietin Stimulating Agents (ESA)
Brief Title: Canakinumab With Darbepoetin Alfa in PTs With Lower-Risk MDS Who Have Failed ESA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20552; CACZ885TUS02T (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — canakinumab; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1b: Dose Level 1 (Experimental): Patients will be treated at dose level 1: Canakinumab 150 mg by subcutaneous injection on day 1 of each 28 day cycle. Darbepoetin alfa will be administered subcutaneously at a dose of 300mg on days 1 and 15 of each cycle.
  Interventions: Drug: Canakinumab Injection; Drug: Darbepoetin Alfa
- Phase 1b: Dose Level 2 (Experimental): Patients will be treated at dose level 2: Canakinumab 300 mg by subcutaneous injection on day 1 of each 28 day cycle. Darbepoetin alfa will be administered subcutaneously at a dose of 300mg on days 1 and 15 of each cycle.
  Interventions: Drug: Canakinumab Injection; Drug: Darbepoetin Alfa
- Phase 2: Treatment at Maximum Tolerated Dose (Experimental): Patients will be treated with Darbepoetin alfa subcutaneously at a dose of 300 mg on days 1 and 15 of each cycle plus the maximum tolerated dose of Canakinumab.
  Interventions: Drug: Canakinumab Injection; Drug: Darbepoetin Alfa

INTERVENTIONS:
Drug: Canakinumab Injection — Participants will be treated at 1 of 2 dose levels of Canakinumab, beginning at 150 mg and increasing to 300 mg or the Maximum Tolerated Dose
  Other Names: Ilaris
Drug: Darbepoetin Alfa — Participants will receive Darbepoetin alfa subcutaneously at a dose of 300mg on days 1 and 15 of each cycle
  Other Names: Aranesp

SUMMARY:
This study is a multi-institution, open-label, Phase 1b/2 clinical trial evaluating the toxicity and efficacy of canakinumab in combination with darbepoetin alfa in patients with lower-risk MDS who have failed prior treatment with an Erythropoietin Stimulating Agent (ESA)

DETAILED DESCRIPTION:
This study is a multi-institution, open-label, Phase 1b/2 clinical trial evaluating the toxicity and efficacy of canakinumab in combination with darbepoetin alfa in patients with lower-risk MDS who have failed prior treatment with an ESA. The study will be conducted in two parts, an initial Phase 1b dose escalation study followed by a dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Adequate organ function as defined by laboratory values per protocol
* Documented diagnosis of MDS by World Health Organization (WHO) criteria, further meeting the following criteria according to disease risk classification
* Patients must be transfusion dependent, defined as requirement for transfusion of at least 3 units of Packed Red Blood cells (PRBCs) 16 weeks for a Hgb<9.0g/dL or, in non-transfusion dependent patients (<3 units of PRBCs transfused in the preceding 16 weeks), must have a baseline Hgb of <9.0 g/dL at time of study enrollment
* Eastern Cooperative Oncology Group (ECOG) Performance Status </=2.
* Women of child bearing potential must have negative urine or serum pregnancy test within 28 days prior to start of study drug.
* Women of child bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence; tubal ligation, partner's vasectomy) prior to Cycle 1 Day 1 and for the duration of study participation.

Exclusion Criteria:

* Use of chemotherapeutic agents or experimental agents (agents that are not commercially available) for the treatment of MDS within 14 days of the first day of study drug treatment.
* Previous treatment with a hypomethylating agent (such as azacitidine, decitabine or investigational hypomethylating agent).
* Use of concurrent growth factors such as G-CSF, GM-CSF, or thrombopoietin mimetics during study except in cases of febrile neutropenia, where G-CSF can be used for short term. Growth factors must be stopped two weeks prior to study.
* Patient has any of the following cardiac abnormalities: (a) Uncontrolled, symptomatic congestive heart failure as designated by the treating physician (b) Myocardial infarction ≤ 6 months prior to enrollment (c) Unstable angina pectoris as designated by the treating physician (d) Serious uncontrolled cardiac arrhythmia as designated by the treating physician. (e) Uncontrolled hypertension as designated by the treating physician
* Known history of human immunodeficiency virus (HIV) (no laboratory testing is required), or active infection with Hepatitis B or Hepatitis C.
* Active tuberculosis (Tb) infection or documented, untreated latent Tb infection (all patients should undergo Tb risk evaluation prior to enrollment with Tb screening performed as per local guidelines,
* Active, uncontrolled infection at the time of enrollment, except in cases of localized infections that are unlikely to lead to a systemic infection such as onychomycoses or dental caries. Patients with new fever (> 38.0 C) or respiratory symptoms are required to undergo laboratory screening for COVID-19
* Have undergone prior allo-HSCT for the treatment of MDS, or other hematologic disorder, or prior solid organ transplant.
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
* Patients with a condition requiring systemic treatment with corticosteroids within 14 days of study drug administration (i.e. prednisone at doses of >10mg). Inhaled or topical steroids and adrenal/pituitary replacement doses >10mg daily prednisone equivalents are permitted.
* Patients undergoing concurrent treatment with agents targeting tumor necrosis factor alpha (TNF) or IL-1 within 28 days of study enrollment.
* Patients who have received a live-virus vaccine within 30 days before study drug administration (patients should not be treated with live-virus vaccine while undergoing therapy).
* History of allergy or hypersensitivity to either darbepoetin alfa or the study drug or its components.
* Women of child bearing potential who are pregnant or breastfeeding.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Maximum Tolerated Dose (MTD) | up to 28 days per cohort
  Maximum tolerated Dose will be determined by testing increasing doses of canakinumab along with a fixed dose of darbepoetin alfa. Patients will be followed for at least 1 cycle before the safety of each cohort can be fully assessed and decisions made for dose escalation in the next cohort. The MTD is defined as the dose level below which DLT is manifested in ≥33% of the patients or at dose level 2 if DLT is manifested in <33% of the patients (with at 6 patients treated at the MTD).
Phase 2: Rate of Hematologic Improvement-Erythroid (HI-E) response | 8 - 12 weeks from baseline
  To determine the rate of hematologic improvement-erythroid (HI-E) response, defined as red blood cell transfusion independence (RBC-TI) of at least 8 weeks in transfusion dependent patients or a mean Hgb increase of >/=1.5g/dL above baseline sustained for at least 8 weeks in non-transfusion dependent patients.

SECONDARY OUTCOMES:
Phase 1b and Phase 2: Duration of Hematologic Improvement-Erythroid (HI-E) response | Up to 12 months per cohort
  Duration of HI-E response: defined as the total duration for which patient is free from transfusions, or in non-transfusion dependent patients, the duration of sustained Hgb improvement of ./=1.5g/dL above pre-treatment baseline.
Phase 1b and Phase 2: Degree in reduction of PRBC Transfusions | at 24 weeks per cohort
  Degree in reduction of PRBC Transfusions: defined as the total reduction in absolute number of units of PRBCs transfused over the first 24 weeks on study versus the number of units of PRBCs during the 16 weeks prior to treatment
Phase 2: Overall Response Rate (ORR) | Up to 60 months
  Overall Response Rate (ORR) is defined by achieving a complete response (CR), partial response (PR), marrow CR (mCR) or hematologic improvement (HI) by IWG 2006 response criteria in MDS
Phase 2: Duration of Response | Up to 60 months
  Duration of response is defined as the duration that begins on the day patient first achieves a response, until the day that patient loses response/progresses as per IWG criteria or dies.
Phase 2: Overall Survival (OS) | Up to 60 months
  OS is defined as the duration of time starting from first treatment with canakinumab until death
Phase 2: Progression Free Survival (PFS) | Up to 60 months
  PFS is defined as the duration of time starting from first treatment with canakinumab until death or disease progression or transformation, as defined by IWG 2006 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: David A Sallman, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory-Winship Cancer Institute, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE